CLINICAL TRIAL: NCT05696990
Title: 3/7 Resistance Training Method in Cardiac Rehabilitation of Coronary Artery Disease and Heart Failure With Reduced Ejection Fraction
Brief Title: 3/7 Resistance Training Method in Cardiac Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Alexis Gillet, Principal Investigator, Université Libre de Bruxelles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P2020/489
Record Dates: First submitted 2023-01-11; First posted 2023-01-25 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure; Coronary Artery Disease
Keywords: cardiac rehabilitation; resistance training; strength training; exercise for older adults
MeSH Terms: conditions — Heart Failure; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3/7 RT method (Experimental): perform interval- type endurance exercise at high intensity and resistance training with the 3/7 method
  Interventions: Other: 3/7 Resistance Training Method
- 3X9 RT method (Active Comparator): perform interval- type endurance exercise at high intensity and resistance training with the 3X9 method
  Interventions: Other: 3X9 Resistance Training Method

INTERVENTIONS:
Other: 3/7 Resistance Training Method — 3/7 Resistance Training Method
  Arms: 3/7 RT method
Other: 3X9 Resistance Training Method — 3X9 Resistance Training Method
  Arms: 3X9 RT method

SUMMARY:
Aim of the clinical monocentric study is to assess the resistance training exercise intervention in patients with Heart Failure with reduced Ejection Fraction (HFrEF) and coronary artery disease that will best improve peak oxygen uptake (Peak Vo2) and leg strength (assessed Isokinetic). The investigators hypothesize that resistance training exercise with induced a high stress metabolic is more important exercise with induced than a lower stress metabolic.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Coronary artery diseases
* Heart failure with reduced ejection fraction

Exclusion Criteria:

* angina
* acutely decompensated heart failure
* electrocardiographic evidence of ischemia
* significant valvular disease
* orthopedic/neurologic disorders that limited exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Peak VO2 after 3 months | Baseline and 3 months
  Change in Peak oxygen consumption (VO2) after three 3 months intervention
Change in strength knee extensor after 3 months | Baseline and 3 months
  Change in strength knee extensor (60°/sec) after three months intervention

SECONDARY OUTCOMES:
Change in VE/VCO2 slope after 3 months | Baseline and 3 months
  Change in ventilatory efficiency (VE/VCO2) slope at baseline and 3 months intervention
Change in submaximal exercise capacity after 3 months | Baseline and 3 months
  Submaximal exercise capacity will be measured using watts at the first ventilatory threshold (VT1)
Change in workload maximal after 3 months | Baseline and 3 months
  Change in workload max at baseline and 3 months intervention
Change in Body fat after 3 months | Baseline and 3 months
  Change in Body fat at baseline and 3 months intervention
Change in lean mass after 3 months | Baseline and 3 months
  Change in lean mass at baseline and 3 months intervention
Change in leg lean mass after 3 months | Baseline and 3 months
  Change in leg lean mass at baseline and 3 months intervention
Change in bone mass after 3 months | Baseline and 3 months
  Change in bone mass at baseline and 3 months intervention
Change in Visceral adipose tissue after 3 months | Baseline and 3 months
  Change in Visceral adipose tissue measure by Dual-energy X- ray absorptiometry (DEXA) at baseline and 3 months intervention
Change in hand grip force after 3 months | Baseline and 3 months
  Change in hand grip force on non dominant hand at baseline and 3 months intervention
Change in ventilation metaboreflex function after 3 months | Baseline and 3 months
  Change in ventilation during metaboreflex test at baseline and 3 months intervention (Briefly, the subject is asked to exercise with the non-dominant arm by performing two 5 min handgrip manoeu- vres reaching approximately 50% of pre-determined maximal con- traction, in random order, separated by a 30 min interval: one bout with circulatory occlusion during the last 10 s of exercise and the all 3 min recovery phase ('clamp session'). During the clamp session, forearm cuff inflation to 30 mmHg above systolic blood pressure from the last 10 s of exercise till the end of the 3 min recovery phase; after cuff inflation, the subject is instructed to relax. Ergore- ceptor sensitivity is quantified as the percentage of the ventilatory and haemodynamic response to exercise maintained by circulatory occlusion during the third minute compared with the third minute of basal recovery.)
Change in diastolic blood pressure metaboreflex function after 3 months | Baseline and 3 months
  Change in diastolic blood pressure during metaboreflex test at baseline and 3 months intervention
Change in heart rate at rest after 3 months | Baseline and 3 months
  Change in heart rate at baseline and 3 months intervention
Change in resting heart rate variability at rest after 3 months | Baseline and 3 months
  Change in resting heart rate variability at baseline and 3 months intervention
Change 30 s sit-to-stand after 3 months | Baseline and 3 months
  Change 30 s sit-to-stand at baseline and 3 months intervention
Change in isometric strength knee extensor after 3 months | Baseline and 3 months
  Change in strength knee extensor (isometric) at baseline and 3 months intervention
Change in 120°/sec strength knee extensor after 3 months | Baseline and 3 months
  Change in strength knee extensor (120°/sec) at baseline and 3 months intervention
Change in 180°/sec strength knee extensor after 3 months | Baseline and 3 months
  Change in strength knee extensor (180°/sec) at baseline and 3 months intervention
Change strength knee extensor in leg extension after 3 months | Baseline and 3 months
  Change in one repetition maximal in leg extensor machine at baseline and 3 months intervention
Change in sub maximal strength knee extensor in leg extension after 3 months | Baseline and 3 months
  Change in 10 repetitions maximal in leg extensor machine at baseline and 3 months intervention
Change in heart rate recovery after 3 months | Baseline and 3 months
  Change in heart rate recovery at baseline and 3 months intervention

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Gillet, Principal Investigator — Université Libre de Bruxelles
Locations (1):
- Erasme Hospital, Brussels, Belgium

REFERENCES:
- [Background] Stragier S, Baudry S, Carpentier A, Duchateau J. Efficacy of a new strength training design: the 3/7 method. Eur J Appl Physiol. 2019 May;119(5):1093-1104. doi: 10.1007/s00421-019-04099-5. Epub 2019 Feb 12. PMID 30756168
- [Background] Duchateau J, Stragier S, Baudry S, Carpentier A. Strength Training: In Search of Optimal Strategies to Maximize Neuromuscular Performance. Exerc Sport Sci Rev. 2021 Jan;49(1):2-14. doi: 10.1249/JES.0000000000000234. PMID 33044332